CLINICAL TRIAL: NCT00837590
Title: Vascular Function, Endothelin, and Inflammation in Pre-diabetic Obesity Versus Lean Healthy Controls
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preliminary results indicated no measurable benefit.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IU-IRB-0901-03
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2013-05

CONDITIONS: Pre-diabetes; Obesity
Keywords: Vascular function; Glucose tolerance; Obesity; Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acute Salsalate (Experimental): Nondiabetic lean and obese subjects will be studied in this arm. Subjects will be studied at baseline and after a single dose of oral salsalate.
  Interventions: Drug: Acute Salsalate
- Chronic Salsalate - Obese (Experimental): Obese subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months' treatment with oral salsalate.
  Interventions: Drug: Chronic salsalate
- Chronic Salsalate - Lean (Experimental): Lean subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months' treatment with oral salsalate. The effects of an acute fatty acid infusion on vascular function will be measured on both occasions.
  Interventions: Drug: Chronic salsalate

INTERVENTIONS:
Drug: Chronic salsalate — Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
  Arms: Chronic Salsalate - Lean; Chronic Salsalate - Obese
Drug: Acute Salsalate — Subjects will receive a single oral dose of 2 gram of oral salsalate
  Arms: Acute Salsalate

SUMMARY:
Aims:

1. Does inflammation contribute importantly to concurrent defects in vascular and metabolic dysfunction in human pre-diabetic obesity?
2. Are there benefits of anti-inflammatory treatment strategies in pre-diabetic obesity in the context of existing treatment with metformin?
3. Are there benefits of anti-inflammatory treatment strategies in pre-diabetic obesity in the context of existing treatment with lisinopril?

DETAILED DESCRIPTION:
We set out to pursue the following Aims:

1. Does inflammation contribute importantly to concurrent defects in vascular and metabolic dysfunction in human pre-diabetic obesity? Pilot studies were performed exploring the acute actions of salsalate on vascular function, the chronic actions of salasate in obese individuals, and actions of chronic salsalate to prevent vascular dysfunction induced by fatty acids in lean individuals.
2. Are there benefits of anti-inflammatory treatment strategies in pre-diabetic obesity in the context of existing treatment with metformin? No studies were performed
3. Are there benefits of anti-inflammatory treatment strategies in pre-diabetic obesity in the context of existing treatment with lisinopril? No studies were performed

The intent of the current project is to efficiently and at low cost generate preliminary data along each of these lines of questioning, studying the minimum number of subjects required to assess the viability of the question using the current measurement approaches.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normotensive (BP<140/95 mmHg)
* lean and obese
* 18 and 55 years
* women must be premenopausal

Exclusion Criteria:

* use of pharmacologic agents or recreational drugs, with the exception of occasional use of non-narcotic pain medications
* blood pressure (>140/90 mmHg)
* elevated cholesterol (LDL >130 mg/dL)
* diabetes mellitus (by ADA criteria)
* evidence of coronary and/or peripheral vascular disease by history and physical exam
* >5 kg change in weight in the preceding 3 months
* chronic systemic illness with recognized metabolic effects
* hepatitis C and HIV
* recognized systemic inflammatory or autoimmune processes such as rheumatoid arthritis or systemic lupus erythematosis
* Raynaud's phenomenon or other abnormalities of hand or finger perfusion
* regular participation in endurance or high-performance athletic activity
* history of aspirin or salsalate sensitivity including aspirin-induced asthma
* prior treatment with salsalate, pentoxyfilline, or monoclonal anti-TNFalpha antibodies
* pregnancy
* liver transaminase levels >3 times the upper limit of normal
* creatinine >1.5 mg/dL
* history of a cellular immunodeficiency-related opportunistic infections, such as an endemic mycosis (eg. histoplasmosis) or mycobacterial infection (eg tuberculosis)
* reactive tuberculin skin test
* history of malignancy except for basal cell carcinoma of the skin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kieren J Mather, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana Clinical Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were self-referred to the clinic for this study.
Pre-assignment Details: Subjects were excluded primarily for anemia based on screening labs or failure to return for clinic visits.
Groups:
- Acute Salsalate: Nondiabetic lean and obese subjects will be studied in this arm. Subjects will be studied at after a single oral dose of salsalate
- Chronic Salsalate - Obese: Obese subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months of treatment with salsalate.
  salsalate : Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
- Chronic Salsalate - Lean: Lean subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months of treatment with salsalate.
  salsalate : Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
Period: Overall Study
Arm/Group | Acute Salsalate | Chronic Salsalate - Obese | Chronic Salsalate - Lean
Started | 6 | 5 | 5
Completed | 6 | 4 | 4
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Acute Salsalate: Nondiabetic lean and obese subjects will be studied in this arm. Subjects will be studied at baseline and after a single dose of salsalate.
  salsalate : Subjects will receive a single day of 4 gram/day of oral salsalate divided into 3 doses.
- Chronic Salsalate - Lean: Nondiabetic lean subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months of treatment with salsalate.
  Salsalate : Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
- Chronic Salsalate - Obese: Nondiabetic obese subjects will be studied in this arm. Subjects will be studied at baseline and after 2 months of treatment with salsalate.
  Salsalate : Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
- Total: Total of all reporting groups
Arm/Group | Acute Salsalate | Chronic Salsalate - Lean | Chronic Salsalate - Obese | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 5 | 16
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 4 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Vascular Function
Description: The primary endpoints of interest is flow-mediated vasodilation
Time Frame: Measured at baseline and after a single oral dose of salsalate (Acute) or 2 months' treatment with salsalate (Chronic)
Population: Pilot study. Analyzing data from all participants completing treatment.
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- Acute Salsalate: Nondiabetic lean and obese subjects will be studied in this arm. Subjects will be studied at baseline and after a single oral dose of salsalate
Arm/Group | Acute Salsalate | Chronic Salsalate - Obese | Chronic Salsalate - Lean
Number analyzed (Participants) | 6 | 5 | 5
ml/min
  Baseline | 5.4 (2.3) | 6.7 (1.7) | 8.3 (2.8)
  Salsalate | 5.6 (1.5) | 4.4 (2.8) | 7.5 (3.9)

ADVERSE EVENTS:
Time Frame: Participants in the Acute protocol participated for two one-day visits approximately 14 days apart. Participants in the Chronic protocols participated for approximately 2 months, with measurements made before and after 2 months of treatment. Total study duration was approximately 17 months from first participant started to final participant completed.
Groups:
- Acute Salsalate: Nondiabetic lean and obese subjects will be studied in this arm. Subjects will be studied before and after a single oral dose of salsalate.
- Chronic Salsalate - Obese: Obese subjects will be studied in this arm. Subjects swill be studied at baseline and after 2 months of treatment with salsalate.
  salsalate : Subjects will receive 2 months of treatment with 4 gram/day of oral salsalate divided into 3 doses.
Arm/Group | Acute Salsalate | Chronic Salsalate - Obese | Chronic Salsalate - Lean
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
This study was a small pilot not powered for main outcomes; the goal was to gather preliminary data for future grants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No